CLINICAL TRIAL: NCT01293955
Title: A Randomized, Double Blinded, Parallel Group, Placebo-controlled Clinical Trial to Assess the Protective Effect of JOINS on Cartilage in Knee Osteoarthritis
Brief Title: Assessment of Protective Effect of JOINS on Cartilage in Knee Osteoarthritis
Acronym: Joins_Carp_Ⅳ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Joins_Carp_IV_2009
Record Dates: First submitted 2010-11-23; First posted 2011-02-11 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Knee Osteoarthritis
Keywords: cartilage; knee osteoarthritis; protective effect
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JOINS 200mg (Experimental): One tablet of JOINS 200mg is administered three times a day for 1 year. The subjects who consent to participate in an extension study are treated with JOINS 200mg for another 1 year.
  Interventions: Drug: JOINS 200mg
- Placebo (Placebo Comparator): One tablet of Placebo is administered three times a day for 1 year. The subjects who consent to participate in an extension study are treated with Placebo for another 1 year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JOINS 200mg — 1 tablet at each time, 3 times a day
  Other Names: JOINS
  Arms: JOINS 200mg
Drug: Placebo — placebo of Joins 200mg
  Arms: Placebo

SUMMARY:
* A Pilot study
* Randomized and Double-blinded
* Placebo controlled
* In 2 parallel group (JOINS 200mg:Placebo = 1:1)
* Overall 24 months treatment (JOINS:Placebo comparison up to 12 months, Additional follow-up assessment up to 24 months)
* Provide rescue medicine throughout whole clinical trial period.

DETAILED DESCRIPTION:
1. Assessment of Efficacy

   1. Knee MRI(Magnetic resonance imaging):

      * Assessment of cartilage volume, thickness in target knee
      * GAG(glycosaminoglycan) concentration of target knee
      * Assessment of Whole-Organ Magnetic Resonance Imaging Score (WORMS) of target knee
   2. Knee radiography:

      * Assessment of changes in minimal medial JSW(Joint Space Width) of target knee.
   3. Knee pain(VAS)

      * Assessment changes of pain in target knee.
   4. K-WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index for Korean)

      * Assessment score change for pain(5 questions), stiffness(2 questions) and physical function(17 questions).
      * The questionnaire is self-administered by the patients.
   5. Used frequency of rescue medicine.
   6. Biochemical cartilage and bone markers

      * Blood and urine sample will be collected all through the morning after a night fasting period since 10 pm the previous day to avoid the variations.
2. Assessment of Safety

   1. Adverse event
   2. Laboratory assessment
   3. Vital sign
   4. 12-lead ECG
   5. Physical examination
3. Enrollment: 76

ELIGIBILITY:
Inclusion Criteria:

1. A female is eligible if she is of:

   * Non-child bearing potential (i.e., physiologically incapable of becoming pregnant), including any female who is at least 2 year after post- menopausal
   * Child bearing potential and agrees to the acceptable contraceptive methods used consistently and correctly
   * Pregnancy test result of negative at screening
2. Primary Knee OA(Osteoarthritis) on medial femorotibial compartment based on ACR(American College Rheumatology) Criteria.

   * ACR Criteria : With Knee pain and satisfied at least 1 of 3 (① age > 50 years, morning stiffness < 30 minute, ③ Presence of Crepitus and Osteophytes on motion)
3. Appropriately signed and dated informed consent has been obtained

Exclusion Criteria:

1. Rheumatoid arthritis or inflammatory arthritis.
2. Bilateral total knee replacement already treated, or planning for the procedure.
3. Knee prosthesis already implanted, or foreseen within the next year.
4. Clinically significant hip osteoarthritis.
5. Severe renal insufficiency defined as creatinine clearance < 30ml/mln(Cockcroft formula).
6. Clinically significant pulmonary, hepatic, renal or heart disorder or diagnosis crucial disease by investigator ( Glycosuria(Diabetes mellitus) or asthma patients are excluded from this clinical study and the patients who has a clinically significant disease are also excluded.).
7. MRI contraindications : overweight, inferior limb diameter non-fitting the knee antenna, inserted pace-maker, metallic prosthesis( if known to interfere with MRI procedure or if known to be unsafe for MRI), metallic clips, insulin pump, cytostatic pump, hearing aid, essential tremor, claustrophobia, etc,.
8. Allergic reaction to Clinical trial medication.
9. Other clinical trial drugs during the 1 month prior to the screening visit.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Knee MRI | up to 4 times

SECONDARY OUTCOMES:
Knee radiography | up to 4 times
Knee pain(VAS) | up to 6 times
K-WOMAC | up to 6 times
Consumption of rescue medication | up to 6 times
  The quantity of rescue medicine will be counted by investigator and recorded in official clinical research document form.
Biomarker | up to 6 times
  Patients will need to be strictly fasting from the night before the visit. The data of biological cartilage and bone markers will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Myoungchul Lee, PH.D.., Principal Investigator — Orthopedics, Seoul National University hospital
Locations (1):
- Seoul National University hospital, Seoul, South Korea